CLINICAL TRIAL: NCT04265170
Title: A Multicentre Pilot Clinical Trial, Evaluating Blast-X® in Combination With Negative Pressure Wound Therapy (NPWT, VAC®) in Validating 4-Week Wound Area Reduction and Reducing Bacterial Bioburden in Chronic Pressure Ulcers
Brief Title: Evaluating Blast-X® in Combination With Negative Pressure Wound Therapy
Acronym: BlastVac-001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SerenaGroup, Inc. (Network)
Collaborators: Next Science TM (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20192645
Record Dates: First submitted 2020-01-28; First posted 2020-02-11 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single-arm (Experimental): Eligible patients are treated with BlastX and VAC. The subjects return to the center three times per week for dressing changes and application of BlastX. The duration of the trial is four weeks and 8 weeks for larger wounds (2 subjects only). Subjects undergo study procedures (biopsy for quantitative tissue culture, photography, fluorescence imaging and swabbing for protease testing) on a weekly basis. The standard of care for pressure ulcers will be continued including debridement, off-loading, and nutritional supplementation when appropriate.
  Interventions: Device: BlastX with negative pressure therapy

INTERVENTIONS:
Device: BlastX with negative pressure therapy — Blast-X in combination with NPWT on,bacterial bio-burden in pressure ulcers assessed by Fluorescence imaging and quantitative biopsy.

SUMMARY:
A Multi-center, Prospective Clinical Trial Evaluating the Combination of BlastX and Negative Pressure Wound Therapy (VAC).To evaluate the 4-week healing trajectory/wound area reduction with BlastX/VAC as compared with historical pre-study 4-week healing trajectory data and data from the US Wound Registry.

DETAILED DESCRIPTION:
The study is a prospective, clinical trial designed to evaluate the combination of BlastX™ and VAC® in facilitating healing and reduction in bio-burden in pressure ulcers. After consenting, the ulcers of eligible subjects are treated with BlastX. After a 5 minute dwell time the wound VAC® is applied as per manufacturers guidelines. The subjects return to the center three times per week for dressing changes and application of BlastX. The duration of the trial is four weeks. Subjects undergo study procedures (biopsy for quantitative tissue culture, photography, fluorescence imaging and swabbing for protease testing) on a weekly basis. The standard of care for pressure ulcers will be continued including debridement, off-loading, and nutritional supplementation when appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with a Full Thickness Pressure Ulcer Stage 3 through Stage 4 without exposed bone of greater than or equal to one month in duration located on the trunk (Sacral, trochanteric, ischial or posterior heel).
2. A signed and dated informed consent form.
3. Subject is able to comply with instructions and scheduled visits.
4. Ulcer surface area >2cm2 and < 100cm2.
5. The patient is a candidate for negative pressure wound therapy.

Exclusion Criteria:

1.Subject or caregiver is unable to manage VAC®device OR the patient cannot return for VAC dressing changes OR the patient does not qualify for home health visits. 2.Subject has major uncontrolled medical disorders such as serious cardiovascular, renal, liver or pulmonary disease, lupus, palliative care or sickle cell anemia.

3.Subject currently being treated for an active malignant disease or subjects with history of malignancy within the wound.

4.The Subject has other concurrent conditions that in the opinion of the Investigator may compromise subject safety.

5.Known contraindications to VAC® or Blast-X® 6.Known allergies to any of the Blast-X®components 7.Concurrent participation in another clinical trial that involves an investigation drug or device that would interfere with this study.

8.Subject is pregnant or breast feeding. 9.Subjects with a history of more than two weeks treatment with immunosuppressants (including systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within one month prior to first Screening Visit, or who receive such medications during the screening period, or who are anticipated to require such medications during the course of the study.

10.Index ulcer has been previously treated with tissue engineered materials (e.g. Apligraf® or Dermagraft®) or other scaffold materials (e.g. Oasis, Matristem) within the last 30 days preceding the first treatment visit.

11.Mini-nutritional assessment Malnutrition Indication score <17. 12.Patient does not have adequate 4-week historical data on comparison in change of wound measurements, photos, costs and supplies used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Wound reduction in surface area | 4 week
  The number of subjects whose wounds reduce in surface area by more than 40% in four weeks

SECONDARY OUTCOMES:
Wounds have a reduction in bacterial load | 4 weeks
  The number of subjects whose wounds have a reduction in bacterial load to below 10^4 as measured by fluorescence imaging
Wounds have a reduction in inflammatory proteases | 4 weeks
  The number of subjects whose wounds have a reduction in inflammatory proteases (matrixmetalloproteases 2,8 and 9 and Human Neutrophil elastase as measured with a standardized point-of-care test
Reduction in wound-related pain | 4 weeks
  The number of subjects who report a reduction in wound-related pain as measured on a Numerical Rating Scale
Incidence of device-related adverse events | 4 weeks
  The incidence of device-related adverse events (Safety and Tolerability)

CONTACTS AND LOCATIONS:
Locations (1):
- Armstrong County Memorial Hospital, Kittanning, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided